CLINICAL TRIAL: NCT02562781
Title: Is Peri-operative Hyperoxemia a Risk Factor for Postoperative Complications? A Randomised, Prospective Study in Patients Undergoing Vascular Surgery
Brief Title: Is Peri-operative Hyperoxemia a Risk Factor for Postoperative Complications?
Acronym: HYPEROXIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ÖrebroU
Record Dates: First submitted 2014-11-15; First posted 2015-09-29 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Vascular Disease
Keywords: postoperative complications; postoperative cognitive dysfunction; oxygen
MeSH Terms: conditions — Vascular Diseases; Postoperative Complications; Postoperative Cognitive Complications | interventions — Oxygen; Air

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplemental Oxygen (Active Comparator): Inspired oxygen fraction > 0.5 and SpO2 = 98-100%
  Interventions: Drug: Oxygen; Other: Air
- Air or supplemental oxygen (Experimental): Air or lowest possible inspired concentration of oxygen to maintain SpO2 > 90%
  Interventions: Drug: Oxygen; Other: Air

INTERVENTIONS:
Drug: Oxygen — Oxygen in sufficient quantity to maintain SpO2 > 98%
  Other Names: Medical oxygen
Other: Air — Supplemental Oxygen in sufficient quantity to maintain SpO2 > 90%
  Other Names: Medical Air

SUMMARY:
Patients undergoing vascular surgery are at a significantly high risk of perioperative cardiovascular, cerebral and renal events compared to those undergoing non-vascular surgery. This could be because of co-morbidities that are common in this patient group. Additionally, smoking, which is common in this population, may be a contributing factor.

Oxygen therapy has been used for decades in order to reduce the risk of myocardial infarction and stroke in patients undergoing vascular surgery and pre-existing co-morbidities in the belief that increased inspired oxygen increases oxygen delivery to tissues, thereby reducing the risk for hypoxia and cell death. However, several studies published recently have questioned the routine use of high inspired oxygen concentration (hyperoxia) to improve oxygen delivery, specifically in the neonatal period but possibly even following myocardial infarction. This could be explained by the fact that increasing inspired concentrations of oxygen cause vasoconstriction in cerebral and coronary arteries, thereby reducing blood flow. Additionally, increased oxygen causes excessive production of reactive oxygen species (ROS), and repercussion injury from oxidative stress. The latter can lead to apoptosis (cell death) in myocardial or cerebral neurons. Despite the high risks of administering oxygen when not needed, it is routinely used in hospitals all over the world without a doctors prescription.

This study aims to assess peri-operative complications up to 1 year following vascular surgery in patients randomised to receive high inspired oxygen concentration (endpoint: SpO2 98 - 100%) or minimal inspired O2 concentration (endpoint: SpO2 > 90%).

DETAILED DESCRIPTION:
Oxygen is probably one of the commonest "non-prescription" drug used in the hospital and its advantage in several situations including carbon monoxide poisoning, central hypoxia and prior to planned intubation in an acute situation are today well-established and commonly used. Oxygen has been frowned upon in the resuscitation of newborn babies because of the risk of retrolental hypoplasia, now well accepted and adopted in clinical practice. Oxygen has also been traditionally used to increase oxygen carrying capacity in patients presenting with an acute coronary syndrome (ACS), to reduce surgical site infections (SSI), to ensure adequate oxygen delivery to tissues in unconscious patients, during cardiac surgery and for postoperative management, specifically after major surgery. Thus, deliberate use of high inspiratory oxygen concentrations (e.g., 80% or above) is recommended in the treatment of specific intoxications, such as with carbon monoxide or cyanide, wherein hyperbaric oxygen should also be considered. In addition, a high oxygen fraction has been suggested to prevent adverse outcomes after surgery and anesthesia, including a reduction in wound infections and postoperative nausea and vomiting (PONV). In critically ill patients, oxygen delivery to the tissues is often compromised, and supplemental oxygen (e.g., face mask with 10 L oxygen per min) is commonly administered to patients with pneumonia, sepsis, acute coronary syndrome, or stroke - in fact, it is estimated that oxygen is given during transport in approximately one-third of all ambulance journeys.

Several reports published recently have questioned many of the "routine" uses of oxygen and some evidence even seems to point towards negative outcomes in some of these conditions. Specifically, excessive oxygen is likely to do more harm than good in the neonatal period, following cardio-pulmonary resuscitation and likely following acute myocardial infarction. Prospective, randomised studies on this important use of oxygen in the preoperative string are, however, lacking in the literature and in view of theoretical risks for hyperoxemia to several organs, the routine use of high oxygen fractions during the peri-operative phase can be questioned.

This study aims to assess peri-operative complications up to 1 year following vascular surgery in patients randomised to receive high inspired oxygen concentration (endpoint: SpO2 98 - 100%) or minimal inspired O2 concentration (endpoint: SpO2 > 90%).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective vascular surgery (peripheral or aortic surgery),
* No language or cognitive disability
* Written, informed consent

Exclusion Criteria:

* Patients with COPD/other lung diseases that require preoperative oxygen therapy
* Patients undergoing carotid artery surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-11; Primary Completion 2020-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Composite morbidity | 0 - 1 month postoperatively
  Major complications such as MACE, TIA/stroke/renal insufficiency/POCD etc

SECONDARY OUTCOMES:
Long term outcome (Major complications) | 1 month to 1 year postoperatively
  Major complications
Specific outcomes (Major adverse cardiac events (MACE)) | 0 - 1 year postoperatively
  Major adverse cardiac events (MACE)
Specific outcomes (TIA or stroke) | 0 - 1 year postoperatively
  TIA or stroke
Specific outcomes (renal insufficiency including dialysis or renal failure) | 0 - 1 year postoperatively
  renal insufficiency including dialysis or renal failure

OTHER OUTCOMES:
Complication (Re-operation or bleeding) | 0 - 30 days postoperatively
  Re-operation or bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gupta, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (2):
- Sweden (2):
  - University Hospital, Örebro
  - Örebro University Hospital, Örebro